CLINICAL TRIAL: NCT01790789
Title: Stress Reduction During Primary Adjuvant Chemotherapy for Ovarian Cancer
Brief Title: Stress Reduction in Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-0027; OS12706 (Other: University of Wisconsin Carbone Cancer Center); 2013-0027 (Other: Institutional Review Board); A532800 (Other: UW Madison); SMPH\OBSTET & GYNECOL\OB-GYN (Other: UW Madison); NCI-2013-01401 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2018-02

CONDITIONS: Ovarian, Fallopian, and Primary Peritoneal Cancer

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress reduction program (Experimental)
  Interventions: Behavioral: Daily stress reduction program
- Attention control (Other)
  Interventions: Other: Attention control

INTERVENTIONS:
Behavioral: Daily stress reduction program — Subjects will participate in activities of a daily stress reduction program.
  Arms: Stress reduction program
Other: Attention control — Subjects will receive periodic phone calls to review study protocol and will receive stress reduction program materials at the end of the study.
  Arms: Attention control

SUMMARY:
The purpose of this study is to investigate the effects of a stress reduction program on the quality of life of ovarian cancer patients during primary adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an initial diagnosis of ovarian, fallopian tube or primary peritoneal cancer who completed primary ovarian cancer surgery or 3 cycles of neoadjuvant chemotherapy with interval cytoreductive surgery (ICS).
* Final pathology diagnosis of stage I-IV ovarian, fallopian tube or primary peritoneal cancer with plan to receive primary adjuvant chemotherapy or completion of chemotherapy after ICS.
* Receive chemotherapy at the University of Wisconsin-Madison.
* Subjects must be at least 18 years of age.
* English-speaking
* Subjects must be able to use audio media, and read and understand the study manual.
* ECOG performance status 0-2.
* Subjects must have a phone.

Exclusion Criteria:

* Subjects participating in a meditation practice more than 1 hour per week prior to surgery and/or chemotherapy administration.
* Subjects with recurrent ovarian, fallopian tube or primary peritoneal cancer.
* Subjects with diagnosis of Chronic Fatigue Syndrome (CFS).
* Subjects unable to use audio media due to auditory dysfunction.
* Subjects unable to read written English.
* Subjects who are prisoners or incarcerated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Fatigue | 18 weeks (completion of chemotherapy)
  Fatigue will be measured using the NIH PROMIS Cancer Fatigue survey instrument

SECONDARY OUTCOMES:
Natural Killer Cell Activity | 18 weeks (completion of chemotherapy)
  Cytotoxicity assays will be conducted to determine if the meditation-based intervention results in an increase in the ability of the NK cells to recognize and lyse cancer targets.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rose, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/